CLINICAL TRIAL: NCT00278980
Title: Effect of C-Peptide on Diabetic Peripheral Neuropathy, a 6 Months Randomized Double-Blind, Placebo Controlled, Dose-Finding, Multicenter Study, With Parallel Groups
Brief Title: Effect of C-Peptide on Diabetic Peripheral Neuropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Creative Peptides Sweden Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CPSp201
Record Dates: First submitted 2006-01-12; First posted 2006-01-19 (Estimated); Last update posted 2006-01-19 (Estimated); Status verified 2006-01

CONDITIONS: Diabetes Mellitus, Type 1; Diabetic Polyneuropathy
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetic Neuropathies | interventions — C-Peptide

INTERVENTIONS:
Drug: C-peptide

SUMMARY:
The aim of the study is to investigate the effect of C-peptide administration on nerve function in patients with type 1 diabetes and peripheral sensory neuropathy.

DETAILED DESCRIPTION:
It has been observed that C-peptide administration results in an activation of renal tubular and sciatic endoneural Na/K-ATPase of the rat and stimulation of endothelial nitric oxide synthase. The hypothesis is that C-peptide administration may improve peripheral nerve dysfunction in diabetic neuropathy by increasing nerve blood flow and Na/K-ATPase activity. The purpose of the trial is to investigate the effect of C-peptide administration on diabetic peripheral sensory neuropathy in patients with type 1 diabetes and diabetic neuropathy in the lower extremities.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have a duration of type 1 diabetes of more than 5 yrs
* Subjects who are C-peptide deficient
* Subjects who have diabetic distal symmetric neuropathy, according to the criteria defined at the San Antonio Conference on Diabetic Neuropathy 1988
* Subjects who have measurable action potential in the sural nerves
* Subjects who have reduced nerve conduction velocity in the sural nerves

Exclusion Criteria:

* Subjects who have neuropathy or signs of nerve dysfunction which may be a consequence of factors other than type 1 diabetes
* Subjects who have concomitant medication that may interfere with the peripheral nerve function or measurement thereof
* Subjects who are transplanted (islet cell, kidney or pancreas)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180
Dates: Start 2003-10; Study Completion 2004-12

PRIMARY OUTCOMES:
Change in sensory nerve conduction velocity from baseline to 6 mo of treatment

SECONDARY OUTCOMES:
- Change in quantitative sensory tests and
neurological impairment assessment from baseline to 6 mo of treatment
- Safety and tolerability of C-peptide

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Juntti-Berggren, MD, PhD, Principal Investigator — Karolinska University Hospital Solna, Stockholm, Sweden
Locations (1):
- Karolinska University Hospital Solna, Stockholm, Stockholm County, Sweden